CLINICAL TRIAL: NCT00400972
Title: Comparison of GlideScope Videolaryngoscopy to Direct Laryngoscopy for Nasal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Centre (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R-06-467; HSREB 12719
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2007-09

CONDITIONS: Nasal Intubation
Keywords: GlideScope; videolaryngoscopy; intubation; nasal; nasotracheal; laryngoscopy; anesthesia

INTERVENTIONS:
Device: GlideScope videolaryngoscope

SUMMARY:
The purpose of this study is to determine whether nasal intubation assisted by GlideScope videolaryngoscopy is faster, easier, and less traumatic than nasal intubation with conventional direct laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* any patient who is at least 18 years old
* patient requires nasal intubation for surgical indications
* operator has performed at least 10 prior GlideScope intubations (oral or nasal)

Exclusion Criteria:

* cervical spine abnormalities
* known difficult airway
* requires rapid sequence induction
* any other patient in whom the attending anesthesiologist believes usage of the GlideScope is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
time to intubation

SECONDARY OUTCOMES:
ease of intubation (VAS)
incidence of trauma
number of failures
severity of patient sore throat on post-operative day 1

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Jones, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada